CLINICAL TRIAL: NCT00093652
Title: ZD1839 (IRESSA®) With Oxaliplatin and Radiotherapy for Esophageal Carcinoma. A Phase I/II Study With Biologic Correlates
Brief Title: Oxaliplatin, Gefitinib, and Radiation Therapy in Treating Patients With Locally Advanced or Metastatic Esophageal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Masking: None | Purpose: Treatment
Other Study IDs: I 04603; RPCI-I-04603; ZENECA-IRUSIRES0303
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; recurrent esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; squamous cell carcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Gefitinib; Oxaliplatin; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: gefitinib
Drug: oxaliplatin
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining oxaliplatin and gefitinib with radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of oxaliplatin when given together with gefitinib and radiation therapy and to see how well they work in treating patients with locally advanced or metastatic esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of oxaliplatin when administered with gefitinib and radiotherapy in patients with locally advanced or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus or gastroesophageal junction. (Phase I)
* Determine the response rate in patients treated with this regimen. (Phase II)

Secondary

* Determine time to tumor progression and median survival in patients treated with this regimen.
* Determine quality of life in patients treated with this regimen.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a phase I, open-label, dose-escalation study of oxaliplatin followed by a phase II study.

* Phase I: Patients receive oxaliplatin IV over 2 hours on days 1, 15, and 29. Beginning on day 1, patients undergo radiotherapy once daily, 5 days a week, for 5.5 weeks. Patients also receive oral gefitinib once daily on days 1-365. Treatment continues in the absence of disease progression or unacceptable toxicity Approximately 3-6 weeks after the completion of chemoradiotherapy, patients are evaluated. Some patients undergo surgical resection* and possibly receive a second course of oxaliplatin (IV over 2 hours on days 1, 15, and 29) 4-8 weeks after surgery. If surgery is not indicated, some patients may receive an additional course of oxaliplatin.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin until the maximum tolerated dose is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive oxaliplatin, gefitinib, and radiotherapy as in phase I at the MTD. Some patients then either undergo surgical resection* and/or begin a second course of oxaliplatin as in phase I.

NOTE: *Oral gefitinib is discontinued ≥ 7 days before surgery and is restarted when the patient has recovered.

Quality of life is assessed at baseline, 5-6 weeks, and then every 2-3 months for 1 year.

Patients are followed every 2-3 months for 1 year.

PROJECTED ACCRUAL: Approximately 15-45 patients (3-12 for phase I and 12-33 for phase II) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma or squamous cell carcinoma of the esophagus or gastroesophageal (GE) junction

  * Locally advanced or metastatic disease by clinical staging, including esophagogastroduodenoscopy and esophageal ultrasound

    * Stage T2, N0 disease and beyond
  * Bulk of tumor must be in the esophagus of patients with GE junction tumor

    * Bronchoscopy is required if primary esophageal tumor is < 26 cm from the incisors
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* At least 4 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Granulocyte count ≥ 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin normal
* ALT and AST ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Not specified

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Pulmonary

* No clinically active interstitial lung disease

  * Patients with chronic stable asymptomatic radiographic changes are eligible

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method (including barrier) contraception during and for 3 months after study participation
* No peripheral neuropathy ≥ grade II
* No severe hypersensitivity to gefitinib or any of its excipients
* No history of allergy to platinum-based compounds or antiemetics administered with protocol-directed chemotherapy
* No active or ongoing infection
* No other uncontrolled illness
* No other significant clinical disorder or laboratory finding that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent colony-stimulating factors during course 1 of study therapy

Chemotherapy

* More than 4 weeks since prior chemotherapy

Endocrine therapy

* Concurrent steroid therapy allowed

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior non-approved or investigational drugs
* No concurrent administration of any of the following:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Barbiturates
  * Highly-active antiretroviral therapy (HAART)
  * Hypericum perforatum (St. John's wort)
* No other concurrent investigational agents or therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (phase I)
Response (phase II)

SECONDARY OUTCOMES:
Survival
Quality of life
Safety and toxicity
Immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Javle M, Pande A, Iyer R, Yang G, LeVea C, Wilding G, Black J, Nava H, Nwogu C. Pilot study of gefitinib, oxaliplatin, and radiotherapy for esophageal adenocarcinoma: tissue effect predicts clinical response. Am J Clin Oncol. 2008 Aug;31(4):329-34. doi: 10.1097/COC.0b013e318161dc04. PMID 18845990